CLINICAL TRIAL: NCT03009461
Title: Randomized Trial of Sorafenib Plus Hepatic Arterial Infusion with Oxaliplatin and Fluorouracil Versus Sorafenib for Hepatocellular Carcinoma with Major Portal Vein Tumor Thrombosis
Brief Title: Sorafenib Plus Hepatic Arterial Infusion Versus Sorafenib for HCC with Major Portal Vein Tumor Thrombosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xiaodong Wang, MD, Chief Physician, Associate Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPVTT
Record Dates: First submitted 2017-01-02; First posted 2017-01-04 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2021-10

CONDITIONS: HepatoCellular Carcinoma; Portal Vein Thrombosis
Keywords: Hepatocellular carcinoma; Portal vein tumor thrombosis; Hepatic arterial infusion chemotherapy; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sor-HAIC group (Experimental): 400 mg of sorafenib (consisting of two 200-mg tablets) twice daily. hepatic arterial chemotherapy consisted of infusions of oxaliplatin (35 mg/m2 for 2 hours), followed by 5-fluorouracil (600 mg/m2 for 22 hours) on day1-3 every 4 weeks.
  Interventions: Procedure: HAIC; Drug: Sorafenib
- Sor group (Active Comparator): 400 mg of sorafenib (consisting of two 200-mg tablets) twice daily.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Procedure: HAIC — Intra-arterial chemotherapy consisted of infusions of oxaliplatin (35 mg/m2 for 2 hours), followed by 5-fluorouracil (600 mg/m2 for 22 hours) on day1-3 every 4 weeks. For each cycle, leucovorin calcium 200 mg/m2 was intravenously administered for 2 hours from beginning of 5-fluorouracil infusion.
  Arms: Sor-HAIC group
Drug: Sorafenib — 400 mg of sorafenib (consisting of two 200-mg tablets) twice daily.

SUMMARY:
According to the Barcelona clinic liver cancer (BCLC) staging treatment guideline, sorafenib is recommended for Hepatocellular Carcinoma (HCC) with Portal Vein Tumor Thrombosis (PVTT), but HCC with major PVTT (in the main trunk or 1st-order branches of the portal vein) did not benefit much from sorafenib in previous studies. There is no established standard treatment for HCC patients with major PVTT, the investigators conducted a randomized, phase 2 study to investigate the survival benefit of sorafenib plus Hepatic arterial infusion chemotherapy (HAIC) with Oxaliplatin and Fluorouracil versus sorafenib for Hepatocellular Carcinoma with Major Portal Vein Tumor Thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or clinically confirmed hepatocellular carcinoma.
* HCC with major PVTT (in the main trunk or 1st-order branches of the portal vein)
* Child A class
* Patient's Eastern Cooperative Oncology Group (ECOG) performance status must be =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 90g/L
* Total bilirubin =< 2 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normality
* Creatinine =< 1.5 X institutional upper limit of normal
* Albumin >= 30g/L
* Patient must be able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Patients who have had prior chemotherapy with Oxaliplatin or Fluorouracil or sorafenib.
* Patient who is receiving any other investigational agents
* Patient who have a diagnosis of hepatic encephalopathy
* Patients who have a diagnosis of sclerosing cholangitis.
* Patients who have a diagnosis of Gilbert's disease.
* Patients who have clinical ascites
* Patient must not have any uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled diabetes mellitus and hypertension, or psychiatric illness/social situations that would limit compliance with study requirements
* No other malignancy except localized basal cell or squamous cell skin cancer in the past 5 years
* Patient who is pregnant or lactating
* Patient Allergic to Iodine contrast medium
* Uncontrolled severe coagulation disorders (INR < 1.5 in patients not on warfarin therapy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagai H, Mukozu T, Ogino YU, Matsui D, Matsui T, Wakui N, Momiyama K, Igarashi Y, Sumino Y, Higai K. Sorafenib and hepatic arterial infusion chemotherapy for advanced hepatocellular carcinoma with portal vein tumor thrombus. Anticancer Res. 2015 Apr;35(4):2269-77. PMID 25862889
- [Background] Sumie S, Yamashita F, Ando E, Tanaka M, Yano Y, Fukumori K, Sata M. Interventional radiology for advanced hepatocellular carcinoma: comparison of hepatic artery infusion chemotherapy and transcatheter arterial lipiodol chemoembolization. AJR Am J Roentgenol. 2003 Nov;181(5):1327-34. doi: 10.2214/ajr.181.5.1811327. PMID 14573429
- [Background] Kim HY, Kim JD, Bae SH, Park JY, Han KH, Woo HY, Choi JY, Yoon SK, Jang BK, Hwang JS, Kim SG, Kim YS, Seo YS, Yim HJ, Um SH; Korean Liver Cancer Study Group. A comparative study of high-dose hepatic arterial infusion chemotherapy and transarterial chemoembolization using doxorubicin for intractable, advanced hepatocellular carcinoma. Korean J Hepatol. 2010 Dec;16(4):355-61. doi: 10.3350/kjhep.2010.16.4.355. PMID 21415578
- [Background] Nouso K, Miyahara K, Uchida D, Kuwaki K, Izumi N, Omata M, Ichida T, Kudo M, Ku Y, Kokudo N, Sakamoto M, Nakashima O, Takayama T, Matsui O, Matsuyama Y, Yamamoto K; Liver Cancer Study Group of Japan. Effect of hepatic arterial infusion chemotherapy of 5-fluorouracil and cisplatin for advanced hepatocellular carcinoma in the Nationwide Survey of Primary Liver Cancer in Japan. Br J Cancer. 2013 Oct 1;109(7):1904-7. doi: 10.1038/bjc.2013.542. Epub 2013 Sep 5. PMID 24008659
- [Background] Kingham TP, D'Angelica M, Kemeny NE. Role of intra-arterial hepatic chemotherapy in the treatment of colorectal cancer metastases. J Surg Oncol. 2010 Dec 15;102(8):988-95. doi: 10.1002/jso.21753. PMID 21166003
- [Background] Xing M, Kooby DA, El-Rayes BF, Kokabi N, Camacho JC, Kim HS. Locoregional therapies for metastatic colorectal carcinoma to the liver--an evidence-based review. J Surg Oncol. 2014 Aug;110(2):182-96. doi: 10.1002/jso.23619. Epub 2014 Apr 24. PMID 24760444
- [Background] Cho M, Gong J, Fakih M. The state of regional therapy in the management of metastatic colorectal cancer to the liver. Expert Rev Anticancer Ther. 2016;16(2):229-45. doi: 10.1586/14737140.2016.1129277. Epub 2016 Jan 13. PMID 26652741
- [Background] Konstantinidis IT, Do RK, Gultekin DH, Gonen M, Schwartz LH, Fong Y, Allen PJ, D'Angelica MI, DeMatteo RP, Klimstra DS, Kemeny NE, Jarnagin WR. Regional chemotherapy for unresectable intrahepatic cholangiocarcinoma: a potential role for dynamic magnetic resonance imaging as an imaging biomarker and a survival update from two prospective clinical trials. Ann Surg Oncol. 2014 Aug;21(8):2675-83. doi: 10.1245/s10434-014-3649-y. Epub 2014 Mar 25. PMID 24664624
- [Background] Wang X, Hu J, Cao G, Zhu X, Cui Y, Ji X, Li X, Yang R, Chen H, Xu H, Liu P, Li J, Li J, Hao C, Xing B, Shen L. Phase II Study of Hepatic Arterial Infusion Chemotherapy with Oxaliplatin and 5-Fluorouracil for Advanced Perihilar Cholangiocarcinoma. Radiology. 2017 May;283(2):580-589. doi: 10.1148/radiol.2016160572. Epub 2016 Nov 7. PMID 27820684
- [Background] Katagiri S, Yamamoto M. Multidisciplinary treatments for hepatocellular carcinoma with major portal vein tumor thrombus. Surg Today. 2014 Feb;44(2):219-26. doi: 10.1007/s00595-013-0585-6. Epub 2013 Apr 17. PMID 23591833
- [Background] Nakazawa T, Hidaka H, Shibuya A, Okuwaki Y, Tanaka Y, Takada J, Minamino T, Watanabe M, Kokubu S, Koizumi W. Overall survival in response to sorafenib versus radiotherapy in unresectable hepatocellular carcinoma with major portal vein tumor thrombosis: propensity score analysis. BMC Gastroenterol. 2014 May 3;14:84. doi: 10.1186/1471-230X-14-84. PMID 24886354
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Zhu K, Chen J, Lai L, Meng X, Zhou B, Huang W, Cai M, Shan H. Hepatocellular carcinoma with portal vein tumor thrombus: treatment with transarterial chemoembolization combined with sorafenib--a retrospective controlled study. Radiology. 2014 Jul;272(1):284-93. doi: 10.1148/radiol.14131946. Epub 2014 Apr 6. PMID 24708192
- [Background] Llovet JM, Bustamante J, Castells A, Vilana R, Ayuso Mdel C, Sala M, Bru C, Rodes J, Bruix J. Natural history of untreated nonsurgical hepatocellular carcinoma: rationale for the design and evaluation of therapeutic trials. Hepatology. 1999 Jan;29(1):62-7. doi: 10.1002/hep.510290145. PMID 9862851
- [Background] Zhang ZM, Lai EC, Zhang C, Yu HW, Liu Z, Wan BJ, Liu LM, Tian ZH, Deng H, Sun QH, Chen XP. The strategies for treating primary hepatocellular carcinoma with portal vein tumor thrombus. Int J Surg. 2015 Aug;20:8-16. doi: 10.1016/j.ijsu.2015.05.009. Epub 2015 May 27. PMID 26026424
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Derived] Zheng K, Zhu X, Fu S, Cao G, Li WQ, Xu L, Chen H, Wu D, Yang R, Wang K, Liu W, Wang H, Bao Q, Liu M, Hao C, Shen L, Xing B, Wang X. Sorafenib Plus Hepatic Arterial Infusion Chemotherapy versus Sorafenib for Hepatocellular Carcinoma with Major Portal Vein Tumor Thrombosis: A Randomized Trial. Radiology. 2022 May;303(2):455-464. doi: 10.1148/radiol.211545. Epub 2022 Feb 1. PMID 35103539